CLINICAL TRIAL: NCT04276103
Title: Development of a Surgical Assessment Tool for National Policy Monitoring & Evaluation in Ethiopia: A Quality Improvement Study
Brief Title: Surgical Assessment Tool for Ethiopia National Policy Monitoring & Evaluation
Status: Completed | Type: Observational
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: General Electric (Industry); Federal Minstry of Health of Ethiopia (Other Government); Jhpiego (Other)
Responsible Party: Principal Investigator, John Meara, Director Program in Global Surgery and Social Change, Harvard Medical School (HMS and HSDM)
Other Study IDs: IJS-D-19-00363R1
Record Dates: First submitted 2020-01-21; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Global Surgery; Health System; Health Planning; Global Anesthesia; Public Health

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: A baseline assessment of surgical capacity is recommended as a first-step to inform national policy on surgical system strengthening. In Ethiopia, the World Health Organization's Situational Analysis Tool (WHO SAT) was adapted to assess surgical capacity as part of a national initiative: Saving Lives Through Safe Surgery (SaLTS). This study describes the process of adapting this tool and initial results.

Methods: The new tool was used to evaluate fourteen hospitals in the Southern Nations, Nationalities, and People's Region of Ethiopia between February and March 2017. Two analytic methods were employed. To compare this data to international metrics, the WHO Service Availability and Readiness Assessment (SARA) framework was used. To assess congruence with national policy, data was evaluated against Ethiopian SaLTS targets.

ELIGIBILITY:
Inclusion Criteria:

* Fourteen public hospitals (11 primary, 1 general, and 2 specialized) chosen by the regional health bureau
* Hospital staff with willingness to participate in study
* Hospital staff with availability to participate in study

Exclusion Criteria:

* Hospital staff which did not volunteer to participate or refused to participate were excluded.
* Hospital staff not available at the time of visit
* Hospitals not chosen by the regional health bureau

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The Southern Nations, Nationalities and Peoples' (SNNP) Region is one of Ethiopia's eleven regions, occupying the southwest portion of the country. Public hospitals serve the region's population in this area within three tiers - primary, general, and specialized hospitals. An average of four providers were interviewed per facility and participants included hospital leadership (CEOs, medical directors, and matrons), surgeons, integrated emergency surgical officers, obstetrician-gynecologists, mid-level anesthesia providers, and operating room nurses.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-02-23 (Actual); Study Completion 2019-02-23 (Actual)

PRIMARY OUTCOMES:
General service readiness | Cross-Sectional, assesses availability of this infrastructure within the past year in general
  Measured by the number of hospital beds, major operating rooms, surgical/anesthesia/and obstetric providers, and basic infrastructure availability
Basic surgery readiness | Cross-Sectional, assesses availability of tracer items within the past year in general
  Readiness for surgical services was assessed based on the presence of tracer items identified by WHO/USAID Service Availability and Readiness Assessment (SARA) as particularly important for providing basic surgical services. The service specific readiness score is defined as the mean availability of service specific tracer items in three domains (staff and training, equipment, and medicines and commodities).
Comprehensive surgery readiness | Cross-Sectional, assesses availability of tracer items within the past year in general
  Readiness for surgical services was assessed based on the presence of additional tracer items identified by WHO/USAID Service Availability and Readiness Assessment (SARA) as necessary to provide comprehensive surgical services, beyond those needed for basic surgery.

CONTACTS AND LOCATIONS:
Overall Officials: John G Meara, MD, DMD, MBA, Principal Investigator — Harvard Medical School & Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: Yes
Raw data from the survey is available in the study and appendices planned for publication. Additionally, the original source data without identification of the specific hospitals, is available upon request with author consensus.
Supporting Information: Study Protocol, CSR
Time Frame: Once the original study is published, de-identified results will be available by request to the authors.
Access Criteria: Original data may be provided upon request to the authors with consensus approval from all co-authors.